CLINICAL TRIAL: NCT04271943
Title: THE EFFECT OF AEROBIC AND GAME BASED EXERCISES ON COGNITIVE FUNCTIONS IN DEMENTIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, guvencetin, physichal therapist MsC, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1170023
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Dementia
Keywords: DEMENTIA; COMPUTER BASED EXERCISE; COGNITIVE EXERCISE
MeSH Terms: conditions — Dementia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMPUTER BASED EXERCISES (Active Comparator)
  Interventions: Behavioral: Computer Based Exercises
- AEROBIC EXERCISES (Active Comparator)
  Interventions: Dietary Supplement: Aerobic Exercises

INTERVENTIONS:
Behavioral: Computer Based Exercises — For 8 weeks 3 days a week for 45 minutes See-ME Virtual Rehabilitation system with the physical therapist will perform cognitive and physical activity exercises
  Arms: COMPUTER BASED EXERCISES
Dietary Supplement: Aerobic Exercises — For 8 weeks 3 days a week exercise bike with 5 min warm-up 35 min constant speed exercise 5 min cooling, a total of 45 min prescribed by the physiotherapist to the maximum heart rate will do aerobic exercise work. Cardiac values will also be monitored throughout the session
  Arms: AEROBIC EXERCISES

SUMMARY:
With the positive contribution of technological developments to living conditions and improvements in health services, the ratio of elderly population to general population is increasing all over the world. Cognitive decline and deterioration are among the most feared in the elderly and have high costs. Dementia is one of the most common diseases of old age. The prevalence of dementia increases in societies where the elderly population increases. At first, while memory is impaired, functions such as attention, language, visuospatial skills, perception and problem solving are impaired. It is estimated that the number of people living with dementia in the world is now 35.6 million, and it will reach 131.5 million by 2050.

Since there is no treatment or effective disease modifying drug to treat the most common types of dementia to date, the research should focus on the development and implementation of non-pharmacological interventions as an alternative or as an additional treatment. In the field of rehabilitation; regular physical exercises, such as walking, strength and balance exercises, dance and chair exercises, can improve physical and cognitive functions such as fitness, daily functions, executive functions, language and working memory in people living with dementia. Movement activation groups such as psychomotor group therapy have been found to have a positive effect on the social behavior of people living with emotional and dementia. Recent meta-analyzes have shown that physical exercise can help maintain and even improve cognitive function in healthy elderly adults. There is evidence that exercise increases the volume of the prefrontal cortex and anterior hippocampus and may increase neurogenesis.

Computer-based cognitive education has received great attention as a safe, relatively inexpensive and scalable intervention aimed at protecting cognition in older adults. It is an innovative way of exercising in a virtual reality or gaming environment that can help dementia patients to be physically active while being cognitively stimulated.

In our study, it was seen that the number of studies on this subject is small and the devices used in the studies were made with game consoles and there were problems in working with game consoles in patients with dementia. Within the framework of all this information, we aimed to investigate the cognitive effects of physical activity and their differences according to each other with computer assisted exergame study written for rehabilitation in demented individuals; We aim to increase cognitive functions and increase quality of life and reaction time of exergamine dementia.

DETAILED DESCRIPTION:
With the positive contribution of technological developments to living conditions and improvements in health services, the ratio of elderly population to general population is increasing all over the world. The slowdown in the process speed, which also explains the slowdown in learning speed in geriatric individuals, is the modality most affected by aging. It has been reported that cognitive speed decreased by 20% at the age of 40 and by 40-60% at the age of 80. Motor speed also decreases with aging. Cognitive decline and deterioration are among the most feared in the elderly.

Dementia is one of the most common diseases of old age. The prevalence of dementia increases in societies where the elderly population increases. At first, while memory is impaired, functions such as attention, language, visuospatial skills, perception and problem solving are impaired. Attention is the first non-memory cognitive domain affected by dementia. Personality changes, behavior and psychiatric symptoms, physical activity problems, vestibular balance and gait problems are added to the table. Although data on the prevalence of dementia are variable, studies are consistent in showing that the prevalence of elderly disease is increasing. It is estimated that the number of people living with dementia in the world is now 35.6 million, and it will reach 131.5 million by 2050.

Since there is no treatment or effective disease modifying drug to treat the most common types of dementia to date, the research should focus on the development and implementation of non-pharmacological interventions as an alternative or as an additional treatment. Non-pharmacological interventions represent an important complement to standard pharmacological treatment in dementia. Cognitive, physical and psychosocial rehabilitation can improve global function, mental status, and quality of life. These interventions can further reduce social costs. Different approaches such as cognitive rehabilitation, occupational therapy, physical activity, music therapy, art therapy and other interventions have been proposed. Interventions that reach patients before they can be diagnosed with dementia can have the greatest impact. Therefore, it is desirable to develop interventions that are moderate, perhaps diagnosed with mild cognitive impairment, or that target those known at risk.

In the field of rehabilitation; regular physical exercises, such as walking, strength and balance exercises can improve physical and cognitive functions such as daily and executive functions, language and working memory in people living with dementia. Movement activation groups such as psychomotor group therapy have been found to have a positive effect on the social behavior of people living with emotional and dementia. Recent meta-analyzes have shown that physical exercise can help maintain and even improve cognitive function in healthy elderly adults. There is evidence that exercise increases the volume of the prefrontal cortex and anterior hippocampus and may increase neurogenesis.

Since there is no effective treatment for dementia, early diagnosis of symptoms and identification of methods that slow down the progression of the disease have been the main focus of relevant medical research in recent years. While treatments remain unclear, older adults and families are seeking accessible, affordable and effective ways to prevent or improve mild cognitive impairment (MCI). Exergame is a unique form of dual task training that combines physical exercise with cognitive compelling tasks in an interactive game-based way. Unlike the more traditional motor-cognitive dual task exercises that combine different training tasks, the preliminary examination typically involves cognitive challenges directly placed in physical body movements that must be performed to complete the game tasks projected on a screen. Since Exergame is a convenient, relatively safe and fun way to be physically active, it is expected that it will positively affect any negative subjective norms related to exercise.

Computer-based cognitive education has received great attention as a safe, relatively inexpensive and scalable intervention aimed at protecting cognition in older adults. It is an innovative way of exercising in a virtual reality or game environment that can help dementia patients to be physically active while being cognitively stimulated.

It was seen that the number of studies on this subject is small and the devices used in the studies were made with game consoles and there were problems in working with game consoles in patients with dementia. Within the framework of all this information, we aimed to investigate the cognitive effects of physical activity and their differences according to each other with computer assisted exergame study written for rehabilitation in demented individuals; We aim to increase cognitive functions and increase quality of life and reaction time of exergamine dementia individuals.

The study is planned to be carried out in a special care center between April 2019 and May 2020 with the patients who are between the ages of 11-25 and the Mini Mental State Scale (MMSE) aged 65 and over.

Inclusion Criteria:

* 65 years or older and MMSE scale between 11-25
* No traumatic brain injury or stroke history

Exclusion Criteria:

* Cooperation problem
* Unstable or severe medical condition,
* Presence of Bipolar Disorder or Psychotic Disorder
* Any co-morbidity that prevents exercise.

The study was planned as a randomized controlled clinical trial; The cases will be divided into two groups by simple randomization method. The sample size of the study is planned to be 15 for each group and the total number of cases is 30.

TREATMENT PROTOCOL The patients included in the treatment will be divided into two groups that we formed as a result of simple randomization.

Group 1 - Study group: 8 weeks, 3 days a week for 45 minutes See-ME Virtual Rehabilitation system with the physical therapist will perform cognitive and physical activity exercises.

Group 2: Control group: will exercise aerobic exercise prescribed according to maximum heart rate for a total of 45 minutes with a 5 minute warm-up and 35 minutes constant speed exercise for 5 minutes with exercise bike for 3 weeks a week for 8 weeks. Cardiac values will also be monitored throughout the session.

Evaluations of both groups will be made and analyzed at the beginning of the treatment, at the end of the 4th week and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 65 YEARS OLD OR OLDER PEPOPLE WITH DEMENTIA
* BETWEEN 11-25 MINI-MENTAL STATE EXAMINITATION SCORE

Exclusion Criteria:

* COOPERATION PROBLEM
* UNSTABLE MEDICAL CONDITION
* PRESENCE OF BIPOLAR DISORDER OR PSYCHOTIC DISORDER
* ANY CO-MORBIDITY THAT PREVENTS EXERCISE

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
MONTREAL COGNITIVE ASSESSMENT | 10 MINUTE
  The MoCA is a screening tool for individuals with mild cognitive dysfunction. The test assesses 8 domains of cognitive functioning: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
STROOP TEST | 10 MINUTE
  He Stroop test Is a test that is used in the field of psychology and shows the interference that can occur in a task that requires selective attention to be performed.
  The selective attention is the one that allows us to be able to attend to two different stimuli at the same time to carry out an action and to discriminate between them to react to what we consider important.

SECONDARY OUTCOMES:
NOTTINGHAM HEALTH PROFILE | 5 MINUTE
  Generic health-related quality of life measure. The instrument is used to evaluate perceived distress across various populations.
DIGIT SPAN TEST | 5 MINUTE
  The Digit Sequencing Test, alternatively called the Digit Span Test is a key tool for working verbal memory. Usually, the examiner reads a list of numbers as the digit sequencing, and the participant repeats them until an incorrect answer is given. In the Qolty version, an audible module lists the numbers and the examiner inputs them onto the screen module. It can be modulated to digit spans of 1-100 sequences long, with forward and reverse sequencing available as features.

CONTACTS AND LOCATIONS:
Locations (1):
- Guvencetin, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: on 2021